CLINICAL TRIAL: NCT06173180
Title: Clinical Evaluation of Vaginal Suture Knotting Device in the Treatment of Urinary Incontinence in Women
Brief Title: VACS Device Clinical Study for Incontinence Treatment
Acronym: VACS-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soranus ArGe ve Danismanlik Hizmetleri Sanayi Ticaret A.S. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VACS-D 001
Record Dates: First submitted 2023-11-28; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: The participants were randomized into two groups and underwent surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VACS-Minifiks (VACS-D) (Active Comparator): During the surgical procedure, this group operated with VACS-Minifiks.
  Interventions: Device: VACS-D
- Transobturator Tape (TOT) (Active Comparator): During the surgical procedure, this group operated with the commercially available Transobturator Tape (TOT).
  Interventions: Device: TOT

INTERVENTIONS:
Device: TOT — In the Transobturator Tape-TOT operation, the anterior vaginal wall is incised 2 cm sagittal 1.5 cm below the urethra in the dorsal lithotomy position and the paraurethral areas are separated by sharp and blunt dissection and the ischiopubic bone is reached with the finger. The skin is incised so as to remain 1 cm lateral to the ischiopubic ramus on the line passing through the clitoris, and the synthetic tape is placed from outside to inside with special inclined trocars, passing under the urethra close to the medial part of the obturator foramen. Cystoscopy is not performed during the procedure. The vagen mucosa is sutured and the procedure is terminated by inserting a urethral foley catheter. The urethral catheter is removed on postoperative day 1 after the investigator evaluates the patient.
  Arms: Transobturator Tape (TOT)
Device: VACS-D — The VACS-Minifiks procedure is a vaginal application of a natural tissue repair procedure whose efficacy has been proven in the abdominal route. The second difference is that the procedure is performed through a single incision instead of the three incisions used in the Transobturator Tape-TOT operation. Thus, the same goal will be achieved in a less invasive way without placing an artificial permanent implant. There is no difference in parameters such as anesthesia, operation time, and discharge time.
  Arms: VACS-Minifiks (VACS-D)

SUMMARY:
Stress Urinary incontinence (SUI) is a common health condition in the female population. Mid-urethral slings (MUS) have proven to be effective in the treatment of female SUI. Trans-obturator tape (TOT) has been demonstrated to be as effective as retropubic tension-free vaginal tape (TVT) with fewer major complications. In this study, it is aimed to evaluate the effectiveness and safety of a newly developed, innovative medical device, as compared to TOT, in the patients diagnosed with urinary incontinence and requiring the surgical intervention.

DETAILED DESCRIPTION:
The study is an open-label, prospective, parallel-group, randomized, controlled medical device clinical trial, conducted in two centers. The two arms of the trial consist of patients randomized to the new device group and to the TOT group. According to this distribution, one group will be subjected to the operation with the new device, and the other group will be subjected to the operation with a commercially available TOT. Primary objective: Evaluation of the effectiveness of using the new device in the surgical treatment of urinary incontinence. Secondary objectives: Evaluation of the effects of the new device use on patients' quality of life, treatment satisfaction, and sexual functions, as well as assessment of safety. The study includes evaluation of the progress employing objective (pad weight, number of incontinence episodes, urodynamic tests) and subjective tests (questionnaires, diaries) during the 12 months follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Those who have not received radiotherapy
* Women aged 40-65 years
* Accompanying infection according to urine culture results people who do not
* Informed about the study and participated in the study patients who have agreed to participate
* Acceptable contraception during work agree to continue to apply their methods those who
* According to the urodynamic test results, the researcher appropriate to be included in the study by patients with
* After physical and neurological examination inclusion in the study was made by the researcher. eligible patients
* Previous response to standard treatments (medication, etc.) non-responders (non-responders to methods such as pelvic floor muscle exercises (with or without physical therapy), behavioral and lifestyle modifications, continence-assisted pessaries, and pharmacotherapy)

Exclusion Criteria:

* Women who are pregnant, supported by biochemical laboratory findings
* Those in the urinary incontinence category other than SUI
* Those with significant pelvic organ prolapse (e.g., cystocele, rectocele); (as defined by the International Continence Society greater than phase II)
* Those with neurological disorders (e.g., multiple sclerosis, Parkinson's disease)
* Patients with morbid obesity (BMI greater than 40 Those who are)
* Those with abnormal bladder capacity (more than 300 cc large)
* Those with abnormal post-void residuals (50 greater than cc)
* Urethral stricture and bladder neck contracture Those who are
* Spastic bladder
* Those with urinary tract infection (UTI)
* Those with vesicoureteral reflux
* Those with bladder stones
* Those with bladder tumors
* Difficulty understanding and adapting to work is mentally healthy to the extent that it can create patients without
* Fulfill the requirements of the work plan who may have trouble adapting to bring patients
* Negative, as determined by the researcher benefit/risk ratio
* Any research in the previous 30 days treatment (medication or device) has been received.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2022-01-07 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
One-Hour Pad Testing | Baseline, 6 weeks, 3 months, 6 months, 12 months
  This test is performed in a clinical setting. They include a filling phase, during which the patient spends 15 minutes drinking 500 ml of fluid. This is followed by a series of provocative maneuvers, such as coughing and jumping, to try to stimulate urinary leakage. Pads are weighed before and at the end of the test. Pad loss ≥ 2 g is designated as significant or a 'positive pad test.
Twenty-Four-Hour Pad Testing | Baseline, 6 weeks, 3 months, 6 months, 12 months
  This test is performed at home. Women are provided with a set of pads and advised not to modify their normal drinking or activities. The aim of such tests is to document leakage in a normal home environment. Pad loss greater than 4 g is designated as significant or a 'positive pad test'.
Number of Total Daily Incontinence Episodes | 6 weeks, 3 months, 6 months, 12 months
  It was obtained using a three-day bladder diary. Objective. Meaningful for patients. Correlates with patients' daily activities. It may not be directly related to the severity of urine leakage. Subject to variability. Requires patient compliance. Day and night urine leakages were recorded separately by the patient for three days. The mean total score for a day was calculated.
Evaluation of Quality of Life | Baseline, 6 weeks, 12 months
  The Incontinence Quality of Life Scale (I-QOL), consisting of 22 questions, was used to analyze the improvement in quality of life. It is a validated questionnaire. Higher scores indicate a better level of quality of life compared to lower scores.
Urodynamic Assessment | Baseline, 12 months
  The bladder is filled using the catheter and pressure measurements are continuously recorded and patient feedback regarding bladder sensation and urgency. Testing for stress incontinence is performed with coughing and straining. Leak Point Pressure and leakage episodes are recorded and analyzed to provide information regarding the type and severity of incontinence. At the end of the test, urine is passed to assess bladder function further and look for blockage of urinary flow.

SECONDARY OUTCOMES:
Symptomatic Assessment for Overactivitive Bladder | Baseline, 12 months
  Overactive Bladder Assessment Form (OAB-V8), was used for symptomatic evaluation and to assess the impact of symptoms on quality of life. A higher score means a worse outcome. Meaningful for patients. It is standardized. The patient's daily activities are taken into account.
Assess the Impact of the Dysfunction on Quality of Life | Baseline, 12 months
  Urogenital Distress Inventory (UDI-6), was used for symptomatic evaluation and to assess the impact of symptoms on quality of life. A lesser score means a better outcome. Meaningful for patients. It is standardized. The patient's daily activities are taken into account.
Symptomatic Impact Assessment | Baseline, 12 months
  Incontinence Impact Questionnaire (IIQ-7), was used for symptomatic evaluation and to assess the impact of symptoms on quality of life. A lesser score means a better outcome. Meaningful for patients. It is standardized. The patient's daily activities are taken into account. OAB-V8, UDI-6, and IIQ-7 are validated questionnaires and subjective. It was not correlated with the severity of urine leakage.
Assessment of Sexual Function | Baseline, 12 months
  It was used for impact on sexual function using the Female Sexual Function Inventory (FSFI), a validated, gender-specific measure of sexual function.
Assessment of Sexual Function during Intercourse | Baseline, 12 months
  Coital Incontinence Questionnaire (CIQ) is a validated, gender-specific measure of sexual function. It was used for the impact on sexual function during Intercourse.
Post-Voiding Residual (PVR) Urine Volume | Baseline, 12 months
  Volume: Since the device has the potential to affect bladder emptying, measurement of PVR and clinical significance are important. PVR volume will be measured with a catheter as per standardization and an abnormal value above 100 ml will be accepted.
Assessment of Serious Adverse Events and Adverse Events | Intraoperative, postoperative 6 weeks, 3 months, 6 months, 12 months
  Patients will be evaluated for adverse events intraoperatively and at visits.

CONTACTS AND LOCATIONS:
Overall Officials: Cagdas Sahin, Assoc. Prof., Principal Investigator — Ege University Faculty of Medicine Department of Obstetrics and Gynecology; Cenk Yasa, Professor, Principal Investigator — Istanbul Faculty of Medicine, Department of Obstetrics and Gynecology; Ozgur Yeniel, Professor, Study Director — Ege University Faculty of Medicine Department of Obstetrics and Gynecology
Locations (2):
- Turkey (Türkiye) (2):
  - Department of Gynecology and Obstetrics, Department of Surgical Medical Sciences, Istanbul Faculty of Medicine, Istanbul
  - Ege University Faculty of Medicine, Department of Obstetrics and Gynecology, Izmir